CLINICAL TRIAL: NCT03653247
Title: A Phase 1/2, Open-Label, Multicenter, Single-Arm Study to Assess the Safety, Tolerability, and Efficacy of BIVV003 for Autologous Hematopoietic Stem Cell Transplantation in Patients With Severe Sickle Cell Disease
Brief Title: A Study to Assess the Safety, Tolerability, and Efficacy of BIVV003 for Autologous Hematopoietic Stem Cell Transplantation in Patients With Severe Sickle Cell Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 003SCD101
Record Dates: First submitted 2018-08-10; First posted 2018-08-31 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease
Keywords: Intervention: Genetic: BIVV003; Drug: Busulfan; Biological: Plerixafor; Phase: Phase 1/2
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — plerixafor; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BIVV003 (Experimental): Participants will receive plerixafor as subcutaneous (SQ) administration followed by myeloablative conditioning therapy with intravenous (IV) busulfan. BIVV003 will then be administered as a 1-time IV infusion of autologous Cluster of Differentiation 34 + Hematopoietic Stem/Progenitor Cell (CD34+HSPC) transfected ex vivo with zinc finger nuclease (ZFN) messenger ribonucleic acid (mRNAs) targeting the B-cell lymphoma/leukemia 11A (BCL11A) locus.
  Interventions: Biological: Plerixafor; Drug: Busulfan; Genetic: BIVV003

INTERVENTIONS:
Biological: Plerixafor — Plerixafor subcutaneous injection will be administered prior to apheresis.
Drug: Busulfan — Busulfan IV infusion will be administered as myeloablative conditioning therapy.
Genetic: BIVV003 — BIVV003 will be administered as an IV infusion following myeloablative conditioning with busulfan.
  Other Names: Autologous CD34 + hematopoietic stem cells

SUMMARY:
This is an open label, multicenter, Phase 1/2 study in approximately eight adults with severe Sickle Cell Disease (SCD). The study will evaluate the safety, tolerability, and efficacy of autologous hematopoietic stem cell transplantation using BIVV003.

DETAILED DESCRIPTION:
Subject participation in this study will be approximately 136 weeks. Enrolled subjects will be asked to participate in a separate long-term follow-up study to monitor the safety and efficacy of BIVV003 treatment for a total of 15 years post-transplant.

ELIGIBILITY:
Inclusion Criteria

* Ages 18 to 40
* Confirmation of sickle cell disease (SCD) diagnosis (HbSS or HbS[beta]0 genotype)
* Severe SCD, defined as having 1 or more of the following manifestations: Clinically significant neurologic event (example [e.g.], stroke) or any neurological deficit lasting more than 24 hours; History of 2 or more episodes or Acute Chest Syndrome (ACS) in 2 years prior to informed consent (despite adequate supportive therapies such as asthma therapy); Six or more pain crises per year in 2 years prior to informed consent (requiring intravenous [IV] pain management in the outpatient or inpatient hospital setting); History of 2 or more cases or priapism with participant seeking medical care in the 2-years prior to informed consent; Regular RBC transfusion therapy in the year prior to informed consent (having received 8 or more transfusions to prevent vaso-occlusive clinical complications); and Echocardiographic finding of tricuspid valve regurgitant jet (TRJ) velocity of greater than or equal to 2.5 meter per second (m/s)
* Clinically stable to undergo stem cell mobilization and myeloablative hematopoietic stem cell transplantation (HSCT)
* Adequate physiological function, defined as the following: Karnofsky/Lansky Performance of greater than or equal to 60; Acceptable cardiac function as defined in protocol; Acceptable pulmonary function as defined in protocol; Acceptable renal function as defined in protocol; and Acceptable hepatic function as defined in protocol
* Ability to understand purpose and risks of study, provide Informed Consent Form (ICF) and authorization to use protected health information
* Completion of age-appropriate cancer screening
* Willingness to use double-barrier method of contraception through entire study period (for participants of childbearing potential)
* Willingness to receive blood transfusions
* Willingness to discontinue hydroxyurea (HU) at least 30 days prior to stem cell mobilization through Day 100 post-transplantation

Exclusion Criteria:

* Previous receipt of an autologous or allogeneic HSCT or solid organ transplantation
* Previous treatment with gene therapy
* Current enrollment in an interventional study or having received an investigational drug within 30 days of study enrollment
* Pregnant or breastfeeding female
* Female or male who plans to become pregnant or impregnate a partner, respectively, during the anticipated study period
* Contraindication to plerixafor, apheresis, or busulfan
* Treatment with prohibited medication in previous 30 days
* Known allergy or hypersensitivity to plerixafor, busulfan, or investigational product excipients
* History of active malignancy within past 5 years, any history of hematologic malignancy, or a family history of a cancer predisposition syndrome (without negative result of candidate)
* Current diagnosis of uncontrolled seizures
* History of significant bleeding disorder
* Clinically significant infection
* Any major organ dysfunction involving brain, kidney, liver, lung, or heart (e.g., congestive heart failure, pulmonary hypertension)
* Corrected QT interval of more than 500 millisecond (ms) based on screening electrocardiogram (ECG)
* Positive for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Known to have a gamma-globin variant associated with altered oxygen affinity
* Hereditary persistence of fetal hemoglobin (HPFH) or HbF concentration of more than or equal to 20 percent (%) at screening
* Absolute Neutrophil Count (ANC) of less than or equal to 1,000 per microliter
* Platelet count of less than 100,000 per microliter
* History of platelet alloimmunization (precluding ability to provide transfusion support)
* Extensive Red Blood Cell (RBC) alloimmunization (precluding ability to provide transfusion support)
* Judged unsuitable for participation by investigator and/or sponsor

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who are Alive at Post-transplantation Day 100 | Day 100
  The percentage of participants who are alive at post-transplantation Day 100 will be calculated using the Kaplan-Meier estimate.
Percentage of Participants who are Alive at Post-transplantation Week 52 | Week 52
  The percentage of participants who are alive at post-transplantation Week 52 will be calculated using the Kaplan-Meier estimate.
Percentage of Participants who are Alive at Post-transplantation Week 104 | Week 104
  The percentage of participants who are alive at post-transplantation Week 104 will be calculated using the Kaplan-Meier estimate.
Percentage of Participants With Successful Engraftment | Up to Day 42
  Successful engraftment is defined by absolute neutrophil count (ANC) greater than or equal to >=500 cells/microliter (mL) for 3 consecutive days.
Number of Participants With Adverse Events (AEs) | Up to Week 104
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Number of Participants With Serious Adverse Events (SAEs) | Up to Week 104
  An SAE is any untoward medical occurrence that at any dose: Results in death, in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); however, this does not include an event that, had it occurred in a more severe form, might have caused death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.

SECONDARY OUTCOMES:
CD34 + HSPC Yield from Plerixafor Stem Cell Mobilization | Approximately 12 weeks
Proportion of Participants with Sufficient Stem Cell Mobilization for Rescue Aliquot and BIVV003 Production | Approximately 12 weeks
Yield of Zinc Finger Nuclease (ZFN)-edited Investigational Product | Approximately 12 weeks
Time to Initial Neutrophil Recovery Following BIVV003 Infusion | Up to Week 104
Time to Platelet Recovery Following BIVV003 Infusion | Up to Week 104
Percentage of Participants With Maintenance of Absolute Neutrophil Count (ANC) of >=500/mcL to last Participant Visit | Up to Week 104
  Percentage of participants maintaining ANC of >=500/mcL to last Participant Visit (Week 104) will be calculated.
Percentage of Participants With Maintenance of Platelet count of >=50,000/mcL to last Participant Visit | Up to Week 104
  The percentage of participants attaining a post-transplant platelet count of >=50,000/mcL and maintaining this level through last Participant Visit (Week 104) will be calculated.
Change From Baseline in Peripheral Blood Fetal Hemoglobin (HbF) Levels | Baseline up to Week 104
  Change from baseline in HbF up to Week 104 will be assessed.
Change From Baseline in Peripheral Blood Percent (%)F cells | Baseline up to Week 104
  Change from baseline in %F cells up to Week 104 will be assessed.
Change From Baseline in Peripheral Blood Sickle Hemoglobin (HbS) Levels | Baseline up to Week 104
  Change from baseline in peripheral blood HbS levels up to Week 104 will be assessed.
Change From Baseline in Peripheral blood total hemoglobin (Hb) concentration | Baseline up to Week 104
  Change From baseline in peripheral blood total hemoglobin (Hb) concentration up to week 104 will be assessed.
Change From Baseline in Reticulocyte Count | Baseline up to Week 104
  Change from baseline in reticulocyte count up to Week 104 will be assessed.
Change From Baseline in Lactate Dehydrogenase (LDH) Levels | Baseline up to Week 104
  Change from baseline in LDH levels up to Week 104 will be assessed.
Change From Baseline in Haptoglobin Levels | Baseline up to Week 104
  Change from baseline in haptoglobin levels up to Week 104 will be assessed.
Change From Baseline in Serum Bilirubin Levels | Baseline up to Week 104
  Change from baseline in serum bilirubin levels up to Week 104 will be assessed.
Change From Baseline in Patient-Reported Outcomes Measurement Information System 57 (PROMIS-57) Scale Score | Baseline up to Week 104
  Quality of life (QoL) measures including fatigue will be assessed using PROMIS-57 scale. This is a 57-item questionnaire with 8 questions per domain for assessing physical and mental well-being in participants with SCD. 57 questions are summed into a total score, which is transformed into an age specific normalized t-score with 50 representing normal, and lower scores representing increasing disability.
Number of Participants With Sickle Cell Disease (SCD)-related Clinical Events | Baseline up to Week 104
  Number of participants with SCD-related clinical events (including vaso-occlusive crisis [VOC], pain episodes etc.) will be reported.
Number of SCD Related Clinical Events by Severity | Baseline up to Week 104
  Severity will be categorized by toxicity grade according to CTCAE Version 5.0. AEs not listed in the CTCAE Version 5.0 will be evaluated by: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe or medically significant but not immediately life threatening, Grade 4=Life-threatening consequences; Grade 5=Death.
Participants lymphocyte Counts | At Weeks 13 and 52
  Lymphocyte counts will be measured to assess reconstitution of immune function post-BIVV003 transplantation.
Participants Immunoglobulin levels | At Weeks 13 and 52
  Immunoglobulin levels will be measured to assess reconstitution of immune function post-BIVV003 transplantation.
Number of Red Blood Cell (RBC) Transfusions Received During the Post-transplantation Study Period | Up to Week 104
  The number of RBC transfusions received during the Post-Transplantation study period will be reported.
Total Volume of RBC Transfused | Up to Week 104
  Total volume of RBC transfused during the Post-Transplantation study period will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sangamo Therapeutics
Locations (5):
- United States (5):
  - UCSF Benioff Children's Hospital, Oakland, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Investigational Site Number 101, Bethesda, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brusson M, Miccio A. Genome editing approaches to beta-hemoglobinopathies. Prog Mol Biol Transl Sci. 2021;182:153-183. doi: 10.1016/bs.pmbts.2021.01.025. Epub 2021 Mar 1. PMID 34175041